CLINICAL TRIAL: NCT06489431
Title: Irrisept vs Traditional Antibiotic Irrigation for Virgin Penile Prosthesis Placement: A Prospective Non-inferiority Trial
Brief Title: Irrisept vs Traditional Antibiotic Irrigation for Virgin Penile Prosthesis Placement
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Irrimaxcorp (Unknown); Urological Surgeons of Northern California (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 21120903
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Erectile Dysfunction; Penile Prosthesis; Complications, Infection or Inflammation
Keywords: Inflatable Penile Prosthesis; Irrisept
MeSH Terms: conditions — Erectile Dysfunction; Infections; Inflammation | interventions — Chlorhexidine; Gentamicins; Rifampin

STUDY DESIGN:
Intervention Model Description: Non inferiority trial
Who Masked: Participant
Masking Description: Participants will be aware of the two options, however will be randomly selected to receive only one of the two treatments. Investigators will be aware of the treatment as they are administering it
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Traditional Antibiotic Therapy (Active Comparator): Preoperative antibiotic selection, method or preparation, draping, or technique;. the corpora, scrotum, and reservoir space will be irrigated with traditional antibiotics (rifampin, gentamycin, +/-fluconazole) immediately after the space is created in all cases. An additional scrotal irrigation with traditional antibiotics after all components are placed will be performed, as well. The patients will be followed and monitored for penile prosthesis infection as well as any other surgical complications for 1 year post operatively.
  Interventions: Drug: Gentamicin; Drug: Rifampin
- Irrisept only irrigation (Experimental): Preoperative antibiotic selection, method or preparation, draping, or technique;. the corpora, scrotum, and reservoir space will be irrigated with Irrisept only immediately after the space is created in all cases. An additional scrotal irrigation with Irrisept only after all components are placed will be performed, as well. The patients will be followed and monitored for penile prosthesis infection as well as any other surgical complications for 1 year post operatively.
  Interventions: Drug: Chlorhexidine

INTERVENTIONS:
Drug: Chlorhexidine — Irrisept is a self-contained jet lavage that contains chlorhexidine gluconate (CHG) as a preservative to offer broad-spectrum activity against various microorganisms in the bottled solution
  Other Names: Irrisept
  Arms: Irrisept only irrigation
Drug: Gentamicin — Aminoglycoside antibiotic irrigation
  Other Names: Gentak
  Arms: Traditional Antibiotic Therapy
Drug: Rifampin — Antibacterial known to inhibit DNA-dependent RNA polymerase
  Other Names: rifampicin; Rifadin
  Arms: Traditional Antibiotic Therapy

SUMMARY:
The purpose of this study is to assess whether intraoperative irrigation with Irrisept is not inferior to irrigation with multiple antibiotics during placement of a first time inflatable penile prosthesis device.

DETAILED DESCRIPTION:
To conduct a prospective, randomized, controlled trial of all virgin penile prosthesis implantations with the goal of assessing Irrisept's candidacy as an alternative to traditional antibiotic irrigation (Rifampin, Gentamicin for all patients, with the addition of Amphotericin B if patient has a history of diabetics) during penile prosthesis surgery. The investigators believe that Irrisept provides adequate antibacterial and antifungal coverage to serve as an alternative to traditional antibiotic therapy. Additionally, the investigators believe a cost analysis would support the use of Irrisept in the event that non-inferiority is demonstrated.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria include all men undergoing penile prosthesis (any manufacturer) implantation (inpatient or outpatient)

Exclusion Criteria:

* Exclusion criteria include men who are having revision implant surgeries, men who may require intraoperative complex reconstruction including graft for Peyronie's Disease, and transgender males

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Infection Rate of Patients Receiving Traditional Antibiotic Irrigation vs Irrisept Only | 1-2 years
  All patients will be closely followed with appointments at regular intervals for the first year after surgery to monitor for infections as per usual care

CONTACTS AND LOCATIONS:
Overall Officials: Edward Cherullo, MD, Principal Investigator — Rush University; Laurence Levine, MD, Principal Investigator — Rush University
Locations (3):
- United States (3):
  - Urological Surgeons of Northern California, Mountain View, California
  - Rush University Medical Center, Chicago, Illinois
  - Uropartners Surgery Center, Des Plaines, Illinois

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in IPP placement. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact the noted research team

REFERENCES:
- [Background] Karpman E, Griggs R, Twomey C, Henry GD. Dipping Titan implants in Irrisept solution (0.05% chlorhexidine gluconate) and exposure to various aerobic, anaerobic, and fungal species. J Sex Med. 2023 Jun 28;20(7):1025-1031. doi: 10.1093/jsxmed/qdad055. PMID 37158448
- [Background] O'Donnell JA, Wu M, Cochrane NH, Belay E, Myntti MF, James GA, Ryan SP, Seyler TM. Efficacy of common antiseptic solutions against clinically relevant microorganisms in biofilm. Bone Joint J. 2021 May;103-B(5):908-915. doi: 10.1302/0301-620X.103B5.BJJ-2020-1245.R2. PMID 33934664
- [Background] Markel JF, Bou-Akl T, Dietz P, Afsari AM. The Effect of Different Irrigation Solutions on the Cytotoxicity and Recovery Potential of Human Osteoblast Cells In Vitro. Arthroplast Today. 2021 Jan 19;7:120-125. doi: 10.1016/j.artd.2020.11.004. eCollection 2021 Feb. PMID 33521208
- [Background] O'Donnell JA, Wu M, Cochrane NH, Belay E, Myntti MF, James GA, Ryan SP, Seyler TM. Efficacy of Common Antiseptic Solutions Against Clinically Relevant Planktonic Microorganisms. Orthopedics. 2022 Mar-Apr;45(2):122-127. doi: 10.3928/01477447-20211227-05. Epub 2022 Jan 3. PMID 34978511
- [Background] Siddiqi A, Abdo ZE, Springer BD, Chen AF. Pursuit of the ideal antiseptic irrigation solution in the management of periprosthetic joint infections. J Bone Jt Infect. 2021 May 26;6(6):189-198. doi: 10.5194/jbji-6-189-2021. eCollection 2021. PMID 34109103
- [Background] Kia C, Cusano A, Messina J, Muench LN, Chadayammuri V, McCarthy MB, Umejiego E, Mazzocca AD. Effectiveness of topical adjuvants in reducing biofilm formation on orthopedic implants: an in vitro analysis. J Shoulder Elbow Surg. 2021 Sep;30(9):2177-2183. doi: 10.1016/j.jse.2020.12.009. Epub 2021 Jan 30. PMID 33529773
- [Background] Wosnitzer MS, Greenfield JM. Antibiotic patterns with inflatable penile prosthesis insertion. J Sex Med. 2011 May;8(5):1521-8. doi: 10.1111/j.1743-6109.2011.02207.x. Epub 2011 Feb 24. PMID 21521487
- [Derived] Desouky E, Tsambarlis P, Levine LA. Comparing 0.05% chlorhexidine gluconate monotherapy to conventional antibiotic irrigation in de-novo penile prosthesis implantation: a two-center prospective randomized controlled non-inferiority study (preliminary results). Transl Androl Urol. 2024 Sep 30;13(9):1905-1911. doi: 10.21037/tau-24-278. Epub 2024 Sep 26. PMID 39434728
- See also: irrisept home page — https://www.irrisept.com/